CLINICAL TRIAL: NCT03432377
Title: Coffee Consumption and NASH in the French Population.
Acronym: COCANASH
Status: Completed | Type: Observational
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Dr Hugues Blondon, Head of Hepatogastroenterology Service, Versailles Hospital
Other Study IDs: P16/17_COCANASH; 2016-A01872-49 (Registry Identifier: ID RBC)
Record Dates: First submitted 2018-01-24; First posted 2018-02-14 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Non Alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of our study is to evaluate the effect of coffee consumption on the risk of severe liver fibrosis in French patients with NASH.

ELIGIBILITY:
Inclusion Criteria:

Any newly diagnosed case of NASH histologically proven graded according to SAF criteria

Or Metabolic syndrome defined by the IDF 2005 criteria:

* waist size> 94cm (men) or> 80cm (women)
* and the presence of at least two of the following criteria:

  * blood pressure: Systolic ≥ 130mmHg OR diastolic ≥ 85 mmHg OR antihypertensive treatment
  * Triglycerides ≥ 1.5g / L or lipid-lowering therapy
  * HDL cholesterol <0.4 g / L (men) or <0.5 g / L (women) or lipid-lowering therapy
  * fasting blood glucose:> 1 g / L or type 2 diabetes AND Hepatic steatosis diagnosed on liver imaging And liver fibrosis (diagnosed with a FibroScan> 6 KPa)

Exclusion Criteria:

* Age <18 years
* Viral hepatitis and other chronic liver diseases
* Alcohol consumption> 20g / day for women, 30g / day for men
* Liver biopsy or FibroScan dating more than 6 months before inclusion.
* History of bariatric surgery
* Serious psychiatric pathology (psychosis, dementia, severe depression) and patients under legal protection (tutelage, guardianship)
* Solid cancer or progressive hematology or <2 years (except basal cell carcinoma or localized squamous cell carcinoma)
* Severe and terminal chronic renal insufficiency (estimated GFR <30mL / min)
* Recent myocardial infarction <6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-Alcoholic Steatohepatitis
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
To compare coffee caffeine consumption in NASH patients with early (F1-2) vs advanced (F3-4) liver fibrosis in univariate analysis and after adjustment for potential confounding factors. | Day 0

SECONDARY OUTCOMES:
Evaluation of the correlation between the degree of hepatic fibrosis assessed by elastometry (FibroScan) or the histological stage and the caffeine consumption from coffee in univariate analysis and after adjustment for potential confounding factors. | Day 0
Comparison of the percentage of regular coffee drinkers in NASH patients with early (F1-2) vs advanced (F3-4) liver fibrosis in univariate analysis and after adjustment for potential confounding factors. | Day 0
Comparison of total caffeine consumption from all types of drinks in patients with NASH with early (F1-2) vs advanced (F3-4) liver fibrosis in univariate analysis and after adjustment for potential confounding factors. | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Hugues BLONDON, Department head, Principal Investigator — Versailles Hospital
Locations (16):
- France (16):
  - Centre Hospitalier de Béziers, Béziers
  - Centre hospitalier Métropole Savoie, Chambéry
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Groupe Hospitalier Public Sud Oise, Creil
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Hospitalier de Gonesse, Gonesse
  - Centre Hospitalier de Hyères, Hyères
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Centre Hospitalier de Bretagne Sud, Lorient
  - Hôpital de Melun, Melun
  - Centre hospitalier Annecy Genevois, Metz-Tessy
  - Centre hospitalier Montelimar, Montélimar
  - Hôpital de Diaconesses, Paris
  - Centre Hospitalier de Perpignan, Perpignan
  - Centre Hospitalier de Saint Denis, Saint-Denis
  - Centre Hospitalier de Sens, Sens